CLINICAL TRIAL: NCT07119528
Title: Application-Based Integrated Care Approach for Enhancing the Effect of FARAPULSE™ Pulse Field Ablation in Patients With Atrial Fibrillation: Randomized Control Trial
Brief Title: Application-Based Integrated Care in Patients After Pulse Field Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2025-0698
Record Dates: First submitted 2025-07-21; First posted 2025-08-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation Patients Treated With the FARAPULSE™ PFA System
Keywords: Atrial fibrillation; Pulse field ablation; Integrated care; Application
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App education group (Experimental)
  Interventions: Other: AF application enhancing AF education
- No-App education group (Experimental)
  Interventions: Other: AF application without enhancing AF education and drug adhrence

INTERVENTIONS:
Other: AF application enhancing AF education — This group will use AF-application. The app will include content related to anticoagulation therapy, such as: medication reminders or intake confirmation for anticoagulants, the importance of anticoagulation therapy in stroke prevention, the role of antiarrhythmic and rate-control medications in symptom management, the necessity of controlling risk factors such as hypertension, diabetes, and hyperlipidemia, and quality of life and cognitive function assessments through questionnaires.
  Arms: App education group
Other: AF application without enhancing AF education and drug adhrence — This group will use AF-application. However, this application will not contain materials enhancing AF education and adherence.
  Arms: No-App education group

SUMMARY:
"Atrial fibrillation (AF) is known as the most common sustained arrhythmia observed in clinical situation. Pulse Field Ablation (PFA) is a recently introduced, effective atrial fibrillation (AF) ablation modality. PFA is safe for treating patients with AF. The "MANIFEST-17K" international study showed important safety outcomes in 17,642 AF patients undergoing post-approval PFA, including no significant risk of esophageal damage, with PFA. PFA provides an appealing alternative to cryoablation and radiofrequency ablation, which often cause damage to non-targeted tissues, particularly the esophagus and phrenic nerve.

An integrated care approach including risk factor management might be of benefit to the clinical outcomes of patients with AF. A mobile application-based integrated care approach is also relatively new and can reduce the burden of physicians and nurses. Recent studies showed that an integrated care approach to holistic AF care can improve the outcome of population-based studies. However, the effect of the mobile application-based integrated care approach has not been evaluated in ablation patients.

Dementia, a decline in memory and other cognitive functions leading to disability in daily function is a common and feared geriatric condition. Although catheter ablation is one of the main treatments for AF, whether it can improve cognitive function in patients with AF remains unclear. Multiple observational trials have shown that catheter ablation is also associated with a lower risk of cognitive decline, dementia, and improved cognitive testing that can be explained through a variety of pathways.

FARAPULSE™ PFA is becoming a widely used ablation technique in AF patients, and knowing the effect of an application-based integrated care approach after AF PFA ablation, and the change in cognitive function is novel. The hypothesis of the study is that AF freedom will be improved by using an application-based integrated care approach in AF patients after the FARAPULSE™ PFA. Another hypothesis is that because of the short procedure time of PFA, the cognitive function will be improved after PFA, and further improved using an application-based integrated care approach.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter study including about 10 hospitals in South Korea. Among subjects treated with the FARAPULSE™ PFA system, those signing the informed consent form will be included in the study. Patients will be randomly assigned in a 1:1 ratio, with the use of a Web-based randomization system, to receive either Application-based integrated care (AF-App group, n=250) or locally available care (no-AF-App group, n=250). They will be followed by 3 Months, 6 Months, and 12 Months. The primary endpoint includes AF freedom (the "ablation and drug-free").

The app will include content related to anticoagulation therapy, such as: medication reminders or intake confirmation for anticoagulants, the importance of anticoagulation therapy in stroke prevention, the role of antiarrhythmic and rate-control medications in symptom management, the necessity of controlling risk factors such as hypertension, diabetes, and hyperlipidemia, and quality of life and cognitive function assessments through questionnaires.

Follow-up assessments will be conducted upto 12 months after enrollment. The anticipated enrollment period is 2 years, with a follow-up duration of one year.

Participants will have voluntary access to educational materials in the app. Medication adherence will be encouraged through reminder alarms, while other educational components will not have specific evaluation methods. The study investigator is responsible for developing the medication adherence education app. The app's content is currently being finalized, and development will be completed using research funding after study approval.

Randomization will be conducted using an Excel macro function, assigning participants in a 1:1 ratio. The randomization process will be uploaded to iCReaT, an electronic case report form (eCRF) system, allowing verification at the time of participant registration.

Primary Outcome: AF freedom at 12 months post-index procedure. (the "ablation and drug-free"). AF Freedom defined as: Freedom from recurrence of individual types of AF, or new AFLs or Ats between 3 month and 12-Month follow-up requiring additional ablation or AADs.

Secondary Outcomes: AF burden: average AF amount per day measured using 1-, 3- or 7-day Holter monitoring at baseline (before ablation), 6, 12 months after PFA.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were treated with the FARAPULSE™ PFA for AF as a de novo procedure
2. Subjects who are willing and capable of providing informed consent
3. Subjects who are willing and capable of participating in App-base integrated care Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Subjects with a current interatrial baffle or patch
2. Subjects with a known or suspected atrial myxoma
3. Subjects with myocardial infarction within 14 days prior to enrollment
4. Subjects with a recent (within 30 days prior to enrollment) Cerebral Vascular Accident (CVA)
5. Subjects who do not tolerate anticoagulation therapy
6. Subjects with an active systemic infection *
7. Subjects with a presence of atrial known thrombus *
8. Subjects with a known inability to obtain vascular access
9. Subjects who are pregnant or planning to be pregnant
10. Subjects with atrial fibrillation that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
11. Subjects with any prosthetic heart valve, ring, or repair including balloon aortic valvuloplasty
12. Subjects with a contraindication to an invasive electrophysiology procedure where insertion or manipulation of a catheter in the cardiac chambers is deemed unsafe per physician's medical judgment, such as, but not limited to, a recent previous cardiac surgery (e.g., ventriculotomy or atriotomy, CABG, PTCA/PCI/coronary stent procedure/unstable angina) and/or in patients with congenital heart disease where the underlying abnormality increases the risk of the ablation (e.g., severe rotational anomalies of the heart or great vessels)
13. Subjects with a life expectancy of ≤ 1 year per investigator's opinion
14. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor to determine eligibility.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
AF freedom at 12 months post-index procedure. | average AF amount per day measured using 1-, 3- or 7-day Holter monitoring at baseline (before ablation), 6, 12 months after PFA.
  Freedom from recurrence of individual types of AF, or new AFLs or Ats between 3 month and 12-Month follow-up requiring additional ablation or AADs

SECONDARY OUTCOMES:
Atrial fibrillation (AF) burden | upto 12 month follow-up
  Atrial burden refers to the proportion of time a patient experiences atrial fibrillation (AF) during a defined observation period, often expressed as a percentage. It's a crucial quantitative measure that helps in assessing stroke risk, the efficacy of antiarrhythmic treatments, and the need for oral anticoagulation. AF burden is measured using Holter monitoring (24 to 72 hours or sometimes upto 7 days) at baseline (before ablation), 6, and 12 months after PFA.
time to stroke (ischemic and hemorrhagic) | upto 12 month follow-up
  Secondary end points assessed time to stroke (ischemic and hemorrhagic), measured as the time from randomization to the first occurrence of either of these events.
time to transient ischemic attack (TIA) | upto 12 month follow-up
  Secondary end points assessed time to transient ischemic attack (TIA), measured as the time from randomization to the first occurrence of either of these events.
time to systemic embolism | upto 12 month follow-up
  Secondary end points assessed time to systemic embolism, measured as the time from randomization to the first occurrence of either of these events.
time to major bleeding | upto 12 month follow-up
  Secondary end points assessed time to major bleeding, measured as the time from randomization to the first occurrence of either of these events. Major bleeding was defined according to the criteria of International Society on Thrombosis and Haemostasis (ISTH) as clinically overt bleeding which was fatal or associated with any of the following: (a) a fall in hemoglobin level of 2 g/dL or more or documented transfusion of at least 2 units of packed red blood cells, (b) involvement of a critical anatomical site (intracranial, spinal, ocular, pericardial, articular, intramuscular with compartment syndrome, retroperitoneal).
time to clinically relevant non-major bleeding | upto 12 month follow-up
  Secondary end points assessed time to clinically relevant non-major bleeding, measured as the time from randomization to the first occurrence of either of these events. Clinically relevant non-major bleeding define a bleeding event that is neither a major bleed as defined by the ISTH 1 nor a non-clinically consequential minor bleeding event.
time to hospitalization events | upto 12 month follow-up
  Secondary end points assessed time to hospitalization events, measured as the time from randomization to the first occurrence of either of these events.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No